CLINICAL TRIAL: NCT04094636
Title: Physical Training During Hospital Admission With Community-Acquired Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Camilla Koch Rysoe, Principal investigator, MSc, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAP-EX
Record Dates: First submitted 2019-09-05; First posted 2019-09-19 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Community-acquired Pneumonia
Keywords: Physical training
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention: Control (No Intervention): Control group
- In-bed cycling (Experimental): Supervised in-bed cycling
  Interventions: Behavioral: In-bed cycling
- Exercise booklet (Experimental): Supervised physical training with exercises from exercise booklet
  Interventions: Behavioral: Exercise booklet

INTERVENTIONS:
Behavioral: In-bed cycling — Patients will daily perform 30 min of supervised in-bed cycling
  Arms: In-bed cycling
Behavioral: Exercise booklet — Patients will daily perform 30 min of supervised physical training with exercises from the exercise booklet
  Arms: Exercise booklet

SUMMARY:
The purpose of this study is to assess the effect of standard usual care combined with daily supervised physical training during hospitalization with community-acquired pneumonia (CAP) compared to standard usual care alnone.

DETAILED DESCRIPTION:
Community-acuired pneumonia (CAP) is a leading cause of hospitalization worldwide. Despite increased focus on mobilization, hospitalization is associated with bed rest. Bed rest with low levels of physical activity leads to functional deline as well as increased risk of complications.

This study is a randomized controlled trial, which investigates the effect of standard usual care combined with daily supervised physical training in patients hospitalized with CAP compared to standard usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older admitted to hospital with CAP defined as a new infiltrate on chest X-ray/CT and minimum one of the following symptoms: temperature <35˚C or ≥38˚C, cough, pleuritic chest pain, dyspnea, or focal chest signs on auscultation.
* Patients should have an expected admission length of ≥72 hours.
* Patients should be able to move their legs.

Exclusion Criteria:

* Patients unable to give written consent.
* Hospital admission within the last 14 days.
* Severe immunosuppression (cancer chemotherapy ≤28 days, neutropenia ≤1000 cells/μL, ≥20 mg prednisolone-equivalent/day >14 days or other immunosuppressive drugs, HIV infection, former transplant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From admission until discharge (an average of 5 days)
  Number of stays in hospital

SECONDARY OUTCOMES:
Readmissions Number of readmissions | 3-months from discharge
  Time-to-event within 3-months from discharge
Mortality | 6-months from discharge
  Time-to-event within 6-months from discharge
Changes in total lean mass | Day 1, day 5, discharge, 1- and 3-months from discharge
  Dual-energy x-ray absorptiometry scans
Changes in total fat mass | Day 1, day 5, discharge, 1- and 3-months from discharge
  Dual-energy x-ray absorptiometry scans
Changes in total fat-free mass | Day 1, day 5, discharge, 1- and 3-months from discharge
  Bioelectrical impedance analysis
Health-related quality of life | Day 1, discharge, 1-, 3- and 6-months from discharge
  Scoring from -0.624 to 1.000 on the 5-level EQ-5D version (EQ-5D-5L) questionnaire (Danish version), with higher score indicating better health-related quality of life
Activities of daily living | Day 1, discharge, 1 month from discharge and 3 months from discharge
  Scoring from 0 to 100 on the Barthel Index for Activities of Daily Living (ADL) with higher score indicating greater independence.
Muscle strength | At day 1, day 5, discharge, 1- and 3-months after discharge
  Hand grip strength test
Functional ability | Day 1, day 5, discharge, 1- and 3-months after discharge
  30-sec chair stand test
Systemic inflammation | Daily during admission (day 0 to 5), 1- and 3-months after discharge
  Pro- and anti-inflammatory cytokine concentrations measured in pg/ml (IL-6, IL-8, IL-18, IL-1a, IL-10, TNF-alpha)
Physical activity monitoring | During admission (up to 7 days), 7 days from discharge, 7 days from 1- and 3 months follow-up
  AX3 accelerometers

OTHER OUTCOMES:
Self-reported physical activity (PA) level | Answered on day 1, 1-, 3- and 6 months after discharge
  3 groups of PA level (high, medium, low) are established based on the scoring of the international physical activity questionnaire (IPAQ).
  * High PA level: Vigorous-intensity activity on at least 3 days and accumulating a minimum of 1500 MET-minutes/week OR 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of 3000 MET-minutes/week
  * Medium PA level: 3 or more days of vigorous-activity of at least 20 minutes/day OR 5 or more days of moderate-intensity activity or walking of at least 30 minutes/day OR 5 or more days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving a minimum of 600 MET-min/week.
  * Low PA Level: No activity is reported OR some activity is reported but not enough to meet criteria for high or medium PA level group.
Glucose metabolism | Day 1, 1- and 3-months from discharge
  Blood samples drawn during an oral glucose tolerance test
Scoring on the Charlson Comorbidity Index to predict 10-year survival | Day 1
  Scale ranges from 0 to 33 points to predict he 10-year mortality for patients with a range of comorbid conditions
HbA1c | Day 1, 1- and 3-months after discharge
  To assess the average blood glucose levels over the previous 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Lindegaard, MD, PhD, Study Director — Department of Pulmonary and Infetious Diseases, Nordsjællands Hospital
Locations (1):
- Department of Pulmonary and Infectious Diseases, Nordsjællands Hospital, Hillerød, Denmark

REFERENCES:
- [Derived] Ryrso CK, Faurholt-Jepsen D, Ritz C, Hegelund MH, Dungu AM, Pedersen BK, Krogh-Madsen R, Lindegaard B. Effect of Exercise Training on Prognosis in Community-acquired Pneumonia: A Randomized Controlled Trial. Clin Infect Dis. 2024 Jun 14;78(6):1718-1726. doi: 10.1093/cid/ciae147. PMID 38491965
- [Derived] Ryrso CK, Faurholt-Jepsen D, Ritz C, Pedersen BK, Hegelund MH, Dungu AM, Sejdic A, Lindegaard B, Krogh-Madsen R. The impact of physical training on length of hospital stay and physical function in patients hospitalized with community-acquired pneumonia: protocol for a randomized controlled trial. Trials. 2021 Aug 28;22(1):571. doi: 10.1186/s13063-021-05503-2. PMID 34454594